CLINICAL TRIAL: NCT06581510
Title: Custom-Made Zirconia Crowns and 3D Printed Resin Crowns Versus Ready-Made Zirconia Crowns in Primary Molars: A Randomized Controlled Trial
Brief Title: Custom-Made Zirconia Crowns and 3D-Printed Resin Crowns Versus Ready-Made Zirconia Crowns in Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Fatema usama, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-010
Record Dates: First submitted 2024-08-21; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Dental Crowns
Keywords: pediatric esthetic crowns; posterior esthetic crowns
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Custom-Made Zirconia crowns (Experimental): CAD/CAM zirconia crown customized for each patient
  Interventions: Procedure: esthetic dental crowns
- 3D Printed Resin Crowns (Experimental): Printed resin crowns customized for each patient
  Interventions: Procedure: esthetic dental crowns
- Ready-Made Zirconia Crowns (Experimental): Nuu smile ready made zirconia crown
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: esthetic dental crowns — Minimal Preparation of esthetic dental crown
  Arms: 3D Printed Resin Crowns; Custom-Made Zirconia crowns
Procedure: control group — Nuu smile ready-made zirconia crown with its well-known reduction
  Arms: Ready-Made Zirconia Crowns

SUMMARY:
The main problem introduced in this study is the aggressive reduction needed for ready-made zirconia crowns to be passively fitted. In addition, its relatively expensive cost and wear of the opposing tooth structure. In this study, different crown materials will be introduced, such as customized zirconia crowns and novel 3D printed resin crowns who may offer better adaptability and gingival health and are relatively cost effective. The proposed study will help in increasing studies of different crown materials for primary teeth

DETAILED DESCRIPTION:
According to AAPD, pulpally treated or deep carious primary teeth should be restored with full coverage crowns for protection of the remaining tooth structure and integrity of occlusion. Different crown materials and compositions have been introduced; however, each with their own drawbacks. Stainless steel crowns have remained the gold standard for restoring primary molars, with the advantages of minimal preparation needed and better adaptability of margins due to their burnishing ability. On the other hand, stainless steel crowns suffer from poor aesthetics and gingival health. The aesthetics of pre-veneered stainless-steel crowns improved but were significantly reduced when the veneered surface was chipped, which was a major drawback in the crown; in addition to their decreased strength and durability in comparison to stainless steel crowns. Strip crowns and polycarbonate crowns were also introduced; however, because of their weak bonding capacity, they have poor strength and an uncertain position in the posterior primary teeth. Due to the increase of aesthetic demand in pediatric dentistry, zirconia crowns have been introduced. Zirconia crowns present the highest aesthetics compared to different pediatric crowns and highest strength compared to all ceramic restorations. However, they need very deep subgingival preparation, poor adaptability because it can't be crimped due to poor burnishing ability and relatively expensive.

Recently, new advances in pediatric crowns have been introduced including computerized 3D printed resin or milled zirconia crowns. Those recent advances have promising results in aesthetics and strength in comparison to ready-made zirconia crowns. Ready-made zirconia crowns have been an exceptionally good biocompatible material. One of the main benefits of those crowns is their durability alongside an outstanding aesthetic appearance. Furthermore, because of their extremely polished surface, ready-made zirconia crowns have proved to have less plaque buildup when compared to other materials. However, because they are costly, need extensive sub-gingival tooth reduction, and cause wear of opposing tooth structure, there are several clinical restrictions and drawbacks.

New computer-aided design digital models serve as the foundation for three-dimensional (3D) printing technologies, which are sophisticated manufacturing techniques that generate customized 3D objects automatically. With applications in almost all fields of dentistry, three-dimensional printing fabricates excellent fitted, accurate, and biocompatible crowns that may overcome ready-made zirconia crowns.

On the other hand, currently the zirconia-based CAD/CAM system has the strongest fracture strength of any all-ceramic material and has continuously produced the most accurate, aesthetically pleasing replication of natural dentition.

They've been acknowledged by patients and dentists alike. The zirconia-based CAD/CAM system is recommended for crowns and bridges in natural teeth, implants, and telescopic dentures. Customized zirconia crowns could be an alternative to the drawbacks presented in ready-made zirconia crowns

ELIGIBILITY:
Inclusion Criteria:

* Healthy children within age range of 5-8 years old
* Upper and lower primary second molars
* Vital primary second molars
* Cooperative children Frankl scale 3 (positive) and 4 (definitely positive)

Exclusion Criteria:

* Radiographic radiolucency related to the furcation and periapical area or any evidence of root resorption
* Deep bite
* More than 2 walls lost due to caries
* Presence of parafunctional habits

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Functional, biological , and esthetic performance according to FDI clinical criteria | 3,6,9 months
  FDI World Dental Federation scores from 1-5 (highest score 1 and lowest score 5 )
Measure amount of reduction done after preparation | During procedure
  Using superimposition technique
Measure time taken during preparation | During procedure
  Stopwatch / timer from start of preparation till the end of preparation
Measure amount of bleeding during preparation | immediately after completion of the procedure (after reduction and cementation of dental crown)
  Gravimetric method by weighing pre and post procedure gauze on scale

SECONDARY OUTCOMES:
Patient's satisfaction while restoring primary molars | During procedure
  Wong baker Faces scale ( 0 least indication no pain and 5 highest indicating pain)
Measure cost-effectiveness of each crown material | through study completion, an average of 1 year
  Compare costs between different crown materials

CONTACTS AND LOCATIONS:
Locations (1):
- The British university in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alrashdi M, Ardoin J, Liu JA. Zirconia crowns for children: A systematic review. Int J Paediatr Dent. 2022 Jan;32(1):66-81. doi: 10.1111/ipd.12793. Epub 2021 Apr 25. PMID 33772904
- [Background] Alzanbaqi SD, Alogaiel RM, Alasmari MA, Al Essa AM, Khogeer LN, Alanazi BS, Hawsah ES, Shaikh AM, Ibrahim MS. Zirconia Crowns for Primary Teeth: A Systematic Review and Meta-Analyses. Int J Environ Res Public Health. 2022 Feb 28;19(5):2838. doi: 10.3390/ijerph19052838. PMID 35270531
- [Background] Jain S, Sayed ME, Shetty M, Alqahtani SM, Al Wadei MHD, Gupta SG, Othman AAA, Alshehri AH, Alqarni H, Mobarki AH, Motlaq K, Bakmani HF, Zain AA, Hakami AJ, Sheayria MF. Physical and Mechanical Properties of 3D-Printed Provisional Crowns and Fixed Dental Prosthesis Resins Compared to CAD/CAM Milled and Conventional Provisional Resins: A Systematic Review and Meta-Analysis. Polymers (Basel). 2022 Jun 30;14(13):2691. doi: 10.3390/polym14132691. PMID 35808735
- [Background] Dewan H. Clinical Effectiveness of 3D-Milled and 3D-Printed Zirconia Prosthesis-A Systematic Review and Meta-Analysis. Biomimetics (Basel). 2023 Aug 27;8(5):394. doi: 10.3390/biomimetics8050394. PMID 37754145
- [Background] Sztyler K, Wiglusz RJ, Dobrzynski M. Review on Preformed Crowns in Pediatric Dentistry-The Composition and Application. Materials (Basel). 2022 Mar 11;15(6):2081. doi: 10.3390/ma15062081. PMID 35329535